CLINICAL TRIAL: NCT01503957
Title: Double-blind, Randomized, Placebo-controlled, Crossover Clinical Investigation to Evaluate Safety and Efficacy of Nasya in Reducing Symptoms of Allergic Rhinitis When Applied Before Allergen Challenge
Brief Title: Nasya in Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: InQpharm Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: INQ/023411
Record Dates: First submitted 2011-12-27; First posted 2012-01-04 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Allergic Rhinitis
Keywords: Allergic rhinitis; Allergen; Allergy; Dustmite
MeSH Terms: conditions — Rhinitis, Allergic; Hypersensitivity | interventions — Abortion, Induced

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline solution (Placebo Comparator): Nasal spray
  Interventions: Device: Saline solution
- Nasya (Experimental): Thixotropic nasal spray suspension
  Interventions: Device: Nasya

INTERVENTIONS:
Device: Nasya — Thixotropic nasal spray suspension, 2 sprays in each nostril
  Arms: Nasya
Device: Saline solution — Nasal spray, 2 sprays in each nostril
  Arms: Saline solution

SUMMARY:
The purpose of this study is to evaluate safety and efficacy of Nasya in reducing symptoms of persistent allergic rhinitis when applied before allergen challenge.

ELIGIBILITY:
Inclusion Criteria:

* History of persistent allergic rhinitis due to house dust mite allergy ≥ 2 years
* Written informed consent

Exclusion Criteria:

* Clinically significant disease that could interfere with the evaluation of study medication
* Participation in other studies within the last 4 weeks / during the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Difference in Total Nasal Symptom Score | 75 minutes

SECONDARY OUTCOMES:
Difference in Total Nasal Symptom Score | Up to 240 minutes
Difference in Total Ocular Symptom Score | Up to 240 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Minoo Lenarz, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Campus Charité Mitte Klinik und Poliklinik für Hals-, Nasen-, Ohren- heilkunde Charité - Universitätsmedizin Berlin, Charitéplatz 1, Berlin, State of Berlin, Germany